CLINICAL TRIAL: NCT01299324
Title: Feasibility Study of Retrograde Delivery of Autologous Concentrated Bone Marrow Nucleated Cell Therapy for Patients Diagnosed With Congestive Heart Failure (CHF)
Brief Title: Retrograde Delivery of BMAC (Bone Marrow Aspirate Concentrate) for Congestive Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harvest Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHF2011-1
Record Dates: First submitted 2011-01-10; First posted 2011-02-18 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Congestive Heart Failure
Keywords: CHF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMAC Infusion (Experimental): Infusion of autologous bone marrow aspirate concentrated nucleated sells into the coronary sinus
  Interventions: Device: BMAC infusion
- Control (No Intervention): Standard of care only. No infusion

INTERVENTIONS:
Device: BMAC infusion — Infusion of 60 mL of Bone Marrow Aspirate Concentrate
  Other Names: Coronary infusion of BMAC
  Arms: BMAC Infusion

SUMMARY:
The primary objective of this feasibility study is to provide clinical data to demonstrate the safety and activity of a concentrate of nucleated cells from bone marrow aspirate (BMAC) produced with the Harvest Bone Marrow Aspirate Concentrate System for treating patients diagnosed with congestive heart failure (CHF).

DETAILED DESCRIPTION:
To demonstrate that the infusion of bone marrow nucleated cells into the coronary sinus is safe as assessed by adverse event records.

To assess the effect of the infusion of bone marrow nucleated cells on the clinical course of angina and heart failure as measured by QOL questionnaire, Minnesota Living with Heart Failure, NYHA and CCS classification and SPECT.

To assess the effect of the infusion of bone marrow nucleated cells on heart function as measured by ejection fraction (EF) and left ventricular end-diastolic diameter (LVEDD) by ECHO.

To assess the effect of the infusion of bone marrow nucleated cells on the area of ischemia as measured by myocardial SPECT studies and ECHO.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ability to understand the planned treatment.
* Patients with Congestive Heart Failure
* Left ventricular ejection fraction ≤40% by echocardiogram, per ECHO completed 30 days prior to treatment
* Symptomatic heart failure NYHA class III or IV
* Able to comply with all study-related visits
* Able to tolerate study procedures, including bone marrow aspiration, SPECT,
* Able to give informed Consent
* Negative for HcG with a serum pregnancy test
* Patients with controlled diabetes mellitus (HbA1c < 9.0%)
* Hematocrit ≥ 28.0%, White Blood Cell count ≤ 14,000, Platelet count ≥ 50,000,
* Life expectancy of 6 months or more in the opinion of the investigator
* Patients requiring high dose corticosteroid therapy (more than 7.5 mg/day) with 1 month before the aspiration or 6 months after the infusion.
* Serum bilirubin, ALT, AST ≤2.5 time the upper level of normal.
* Controlled blood pressure (systolic blood pressure ≤140 and a diastolic blood pressure of ≤90 mmHG) and established anti-hypertensive therapy as necessary prior to entry into the study
* Patient has received stable, standard medical therapy for at least one month with no new medications to treat the disease introduced in the last 3 months.
* Pre-existing condition (e.g. thromboembolic risk, diabetes, hypercholesterolemia are adequately controlled in the opinion of the investigator)
* Fertile patients (male and female) must agree to use an appropriate form of contraception while participating in the study.

Exclusion Criteria:

* Female who is pregnant or nursing, or of child bearing potential and is not using a reliable birth control method, or who intend to become pregnant during the tenure of this study.
* History of prior radiation exposure for oncological treatment.
* History of Bone Marrow Disorder (especially NHL, MDS) that prohibit transplantation.
* History of abnormal bleeding or clotting.
* History of Liver Cirrhosis.
* End stage renal disease (Creatinine ≤ 3.0 mg / dl) and/or dialysis
* Acute Myocardial Infarction < 1 week from treatment date.
* Active clinical infection being treated by antibiotics within one week of enrollment
* Inability or unwillingness to comply with the treatment protocol, follow-up, research tests, or give consent.
* Unable to have 250cc bone marrow harvested.
* History of life-threatening arrhythmias, except if an automated implantable cardioverter defibrillator (AICD) is implanted
* Life expectancy <6 months due to concomitant illnesses
* Known cancer and undergoing treatment; chemotherapy and/or radiotherapy
* Patients receiving treatment with hematopoietic growth factors (e.g., EPO, G-CSF)
* Patients who can not stop anticoagulation therapy (warfarin) 72hrs prior to bone marrow aspiration and infusion
* Patients who can not stop anti-platelet therapy (clopidogrel) 7 days prior to bone marrow aspiration and infusion
* History of alcohol consumption exceeding the equivalent of 2 drinks/daily (1 drink = 5oz wine, 12oz of beer, or 1.5oz hard liquor) or illicit drug use within 6 months of screening.
* Patient who will require continuous high dose corticosteroid therapy (more than 7.5mg/day) within 1 month before aspiration or 6 months after injection procedure.
* Body Mass Index (BMI) of 40 kg/m2 or greater
* Patient receiving experimental medication or participating in another clinical study within 30 days of signing the informed consent
* In the opinion of the investigator or the sponsor, the patient is unsuitable for cellular therapy
* Known allergy or sensitivity to contrast agents used in imaging procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 12 Months
  To demonstrate that the infusion of bone marrow nucleated cells into the coronary sinus is safe as assessed by adverse event records.

SECONDARY OUTCOMES:
Assess the effect of the infusion of bone marrow nucleated cells on the clinical course of angina | 12 Months
  To assess the effect of the infusion of bone marrow nucleated cells on the clinical course of angina as measured by QOL questionnaire, Minnesota Living with Heart Failure, NYHA and CCS classification and SPECT.
Assess the effect of the infusion of bone marrow nucleated cells on the clinical course of heart failure | 12 Months
  To assess the effect of the infusion of bone marrow nucleated cells on the clinical course of heart failure as measured by QOL questionnaire, Minnesota Living with Heart Failure, NYHA and CCS classification and SPECT.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Patel, MD, Principal Investigator — University of Utah
Locations (3):
- Rostock University Hospital, Rostock, Germany
- Medanta the Medicity, Gūrgaon, India
- Dept of Cardiology, Clinicas Maison de Sante, Lima, Peru